CLINICAL TRIAL: NCT03903198
Title: Care Pathways of Acute Heart Failure Patients: Impact on In-hospital Mortality. A French National Prospective Survey
Brief Title: Care Pathways of Acute Heart Failure Patients: Impact on In-hospital Mortality.
Status: Completed | Type: Observational
Sponsor: frederic ADNET (Other)
Responsible Party: Sponsor-Investigator, frederic ADNET, MD, PhD, Association pour le Développement de la Recherche et de l'Enseignement en Médecine d'Urgence
Organization: Association pour le Développement de la Recherche et de l'Enseignement en Médecine d'Urgence (Other)
Other Study IDs: 1836586v0
Record Dates: First submitted 2019-03-28; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Acute Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators conducted a prospective observational study to describe the different pre-hospital and in-hospital pathways of patients with acute heart failure (AHF) and their association with in-hospital mortality.

DETAILED DESCRIPTION:
Prospective observational national multicentric study in 26 centres. Between june 2014 and october 2018 The investigators collected data about baseline characteristics, first recourse, in-hospital places of care and places of hospitalizations. Lengths of care and lengths of hospitalization.

Collected data of each patient were reported on a specific assessment tool. The investigators ran a univariate analysis and logistic regression between steps of the care pathway and in-hospital mortality. The main result was validated by an analysis with a propensity score: association between a hospitalization in cardiology and in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to hospital with Acute Heart Failure according to the physician in care

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in 26 french hospitals for Acute Heart Failure
Sampling Method: Non-Probability Sample
Enrollment: 3677 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | Between patient's inclusion in the study and it's hospital discharge, up to one year
  Death of the patient during hospital stay reported by the physician in charge

CONTACTS AND LOCATIONS:
Overall Officials: Frederic ADNET, MD, PhD, Principal Investigator — Association pour le Développement de la Recherche et de l'Enseignement en Médecine d'Urgence

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cowie MR, Anker SD, Cleland JGF, Felker GM, Filippatos G, Jaarsma T, Jourdain P, Knight E, Massie B, Ponikowski P, Lopez-Sendon J. Improving care for patients with acute heart failure: before, during and after hospitalization. ESC Heart Fail. 2014 Dec;1(2):110-145. doi: 10.1002/ehf2.12021. Epub 2015 Jan 21. PMID 28834628
- [Background] Cleland JG, McDonagh T, Rigby AS, Yassin A, Whittaker T, Dargie HJ; National Heart Failure Audit Team for England and Wales. The national heart failure audit for England and Wales 2008-2009. Heart. 2011 Jun;97(11):876-86. doi: 10.1136/hrt.2010.209171. Epub 2010 Dec 20. PMID 21173198
- [Derived] Gorlicki J, Boubaya M, Cottin Y, Angoulvant D, Soulat L, Guinemer S, Bloch-Queyrat C, Deltour S, Lambert Y, Juilliere Y, Adnet F. Patient care pathways in acute heart failure and their impact on in-hospital mortality, a French national prospective survey. Int J Cardiol Heart Vasc. 2019 Dec 5;26:100448. doi: 10.1016/j.ijcha.2019.100448. eCollection 2020 Feb. PMID 31867437